CLINICAL TRIAL: NCT02308670
Title: An Open-label, Prospective, Observational, Single-blinded, Longitudinal, Cross-over Study to Evaluate the Effect of Switching From Daily Injections of 20mg Glatiramer Acetate (GA) to 40mg GA Three Times a Week on Thalamic Pathology in Subjects With Relapsing-remitting Multiple Sclerosis
Brief Title: Evaluate the Effect of Switching From Daily Injections of 20mg Glatiramer Acetate (GA) to 40mg GA Three Times a Week in Subjects With Relapsing-remitting Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Robert Zivadinov, University at Buffalo
Other Study IDs: GA20-40
Record Dates: First submitted 2014-07-23; First posted 2014-12-04 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RRMS changing from 20mg to 40mg GA: Relapsing-remitting Multiple Sclerosis patients who are switching from 20mg of glatiramer acetate (GA) to 40mg. The investigator is not influencing this clinical decision, just measuring its impact using MRI metrics.

SUMMARY:
The primary aim of this study is to observe any changes in MRI in MS patients who have switched from 20mg injections/day to 3 40mg injections/week of glatiramer acetate.

DETAILED DESCRIPTION:
The primary aim of this study is to observe the effect of switching from daily injections of 20mg glatiramer acetate (GA) (20mg/daily) to GA 40mg three times a week (40mg x 3/weekly) on thalamus pathology, as measured by changes in diffusion-tensor imaging (DTI) in patients with relapsing-remitting multiple sclerosis (RRMS). We hypothesize that GA 40mg x 3/weekly will exert similar, if not better effect on prevention of thalamic pathology, as compared to GA 20mg/daily. The secondary objective of this study is to investigate the effect of switching from GA 20mg/daily to GA 40mg x 3/weekly on evolution of microstructural changes in normal appearing white matter (NAWM) and normal appearing gray matter (NAGM), as measured by DTI.

ELIGIBILITY:
Inclusion Criteria:

* MS patients diagnosed with MS according to the McDonald criteria
* MS patients having a relapsing disease course
* Being on GA monotherapy (20mg/daily sc) for at least 12 months prior to the standard of care MRI at the time of switch to GA 40mg x 3/weekly
* Having standard of care 3T MRI scan while on GA 20mg/daily treatment for at least 12-18 months prior to the start day of the of the GA 40mg x 3/weekly and at the time of switch to GA 40mg x 3/weekly Age over 18
* Pass MRI health screening (in case of EGFR <59, the contrast will not be applied)
* None of the exclusion criteria

Exclusion Criteria:

* Patients who had a relapse within 30 days prior to MRI scan date
* Patients who received steroid treatment within 30 days prior to the MRI scan date
* Women who are pregnant, lactating or of childbearing age who do not consent to approved contraceptive use during the study
* MS patients who used other imunomodulatory or immunosuppressant treatment other than GA during the 12 months prior to start of GA 40mg 3/weekly (e.g., IFN-β, mitoxantrone, cyclophosphamide, cladribine, fludarabine, cyclosporine, total body, azathioprine, methotrexate, IVIG, cellcept, natalizumab, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred fifty (150) consecutive RRMS patients who are on treatment with GA 20mg/daily for at least 12 months and who switched to GA 40mg x 3/weekly, because of convenience of application, will be recruited in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Absolute and percent change in thalamus pathology as measured by axial and radial diffusivity using diffusion tensor imaging tract-based spatial statistics | 1 year after enrollment
  The primary endpoint is to explore the effect of GA 40mg x 3/weekly on thalamus pathology, as measured by changes in RD and AD on DTI TBSS in patients with RRMS, as compared to GA 20mg/daily.

SECONDARY OUTCOMES:
Absolute and percent changes in normal-appearing white and grey matter as measured by fractional anisotropy and mean diffusivity using diffusion tensor imaging tract-based spatial statistics. | 1 year after enrollment
  The secondary endpoint is to investigate the effect of GA 40mg x 3/weekly on evolution of microstructural changes in NAWM and NAGM, as measured by FA and MD on DTI global and the TBSS (only NAWM) approaches, as compared to GA 20mg/daily.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD, PhD, Principal Investigator — SUNY University at Buffalo
Locations (1):
- Buffalo Neuroimaging Analysis Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zivadinov R, Bergsland N, Hagemeier J, Tavazzi E, Ramasamy DP, Durfee J, Cherneva M, Carl E, Carl J, Kolb C, Hojnacki D, Weinstock-Guttman B. Effect of switching from glatiramer acetate 20 mg/daily to glatiramer acetate 40 mg three times a week on gray and white matter pathology in subjects with relapsing multiple sclerosis: A longitudinal DTI study. J Neurol Sci. 2018 Apr 15;387:152-156. doi: 10.1016/j.jns.2018.02.023. Epub 2018 Feb 10. PMID 29571854